CLINICAL TRIAL: NCT01341119
Title: Retrospective Analysis of Skin/Soft Tissue Primary NK/T Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Other Study IDs: 2010-11-047
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Extranodal NK/T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
To study clinical features, prognostic factors and treatment outcome and to develop a possible prognostic index in skin/soft tissue primary NK/T cell lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed extranodal NK/T cell lymphoma
* primary site is skin or soft tissue

Exclusion Criteria:

* involvement of upper aerodigestive tract

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-11

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea